CLINICAL TRIAL: NCT01058499
Title: Mindfulness Based Stress Reduction in COPD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Roberto P. Benzo, M.D., Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-008478
Record Dates: First submitted 2010-01-27; First posted 2010-01-28 (Estimated); Last update posted 2016-03-21 (Estimated); Status verified 2016-03

CONDITIONS: Chronic Obstructive Pulmonary Disease; COPD
Keywords: Chronic Obstructive Pulmonary Disease; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MBSR (Experimental)
  Interventions: Behavioral: Mindfulness Based Stress Reduction Program (MBSR)

INTERVENTIONS:
Behavioral: Mindfulness Based Stress Reduction Program (MBSR) — Traditional eight-week MBSR Program.

SUMMARY:
The objective of this study is to test the efficacy of a Mindfulness Based Stress Reduction program in COPD on quality of life, dyspnea, daily physical activity and mindfulness during daily life.

ELIGIBILITY:
Inclusion criteria:

* clinical diagnosis of COPD
* clinically significant dyspnea, as determined by a score of >=2 on the Medical Research Council of Dyspnea Score questionnaire (0-4).

Exclusion criteria:

* patients with a high likelihood of not completing the program (active chemical dependency)
* patients with an inability fo provide good data or to follow commands (neurologic or psychiatric condition).
* poor motivation or lack of interest in program

Ages: 40 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-02; Primary Completion 2010-09 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
We hypothesize that the perception of well being will increase after participants go through the MBSR program for COPD. | Baseline and at eight weeks

SECONDARY OUTCOMES:
Participants in the MBSR for COPD will have an increase in their physical activity level. | Baseline and 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Benzo, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States